CLINICAL TRIAL: NCT06070493
Title: The Effects of Myofascial Release Technique in Patients With Rotator Cuff Injury: A Single-Blind Randomized Controlled Trial
Brief Title: The Effects of Myofascial Release Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Tuğçe Çoban, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-77082166-302.08.01-407339
Record Dates: First submitted 2023-09-19; First posted 2023-10-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Injuries
Keywords: Myofascial Release Therapy; Proprioception; Shoulder Pain; Rotator Cuff Lesions
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: The control group received a classical physiotherapy program including transcutaneous electrical nerve stimulation, hot pack and exercise, while the treatment group received the same classic physiotherapy program along with the myofascial release technique. All treatments were planned for 4 weeks and a total of 10 sessions.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): classical physiotherapy
  Interventions: Other: classic physiotherapy program
- Treatment group (Experimental): classical physiotherapy and myofascial release
  Interventions: Other: classic physiotherapy program; Other: Myofascial release

INTERVENTIONS:
Other: classic physiotherapy program — For individuals of control group, a hot pack was applied to the shoulder area for 15 minutes, while the individuals were in the sitting position. The conventional mode of transcutaneous electrical nerve stimulation was used. Frequency was adjusted in the range of 50-100 Hz, and the amplitude intensity was adjusted between 10-30 milliampere with the intensity of mild tingling without causing any excessive discomfort or contractions. Electrodes were placed at the anterior, posterior, superior, and inferior of the shoulder region. In the exercise program of the patients, joint range of motion exercises, stretching, scapular stabilization, rotator cuff, and shoulder muscle strengthening exercises were given.
Other: Myofascial release — myofascial release technique was applied to the patients in the treatment group besides the control group program. The technique was applied to the lateral neck and shoulder, pectoral region, scapulothoracic area, and arm regions for 5 minutes for optimum benefit.
  Arms: Treatment group

SUMMARY:
This study was planned to investigate the long-term effects of myofascial release technique on proprioception, pain severity, shoulder range of motion, functional level, flexibility, and muscle strength in patients with rotator cuff injury. The study included 29 individuals with partial rotator cuff injury who were randomly divided into two groups. The control group received a classical physiotherapy program including transcutaneous electrical nerve stimulation, hot pack and exercise, while the treatment group received the same classic physiotherapy program along with the myofascial release technique. All treatments were planned for 4 weeks and a total of 10 sessions. Proprioception, pain severity, shoulder range of motion, functional level, flexibility and muscle strength were assessed before and after the treatment.

DETAILED DESCRIPTION:
Rotator cuff injury is the most common cause of shoulder pain and dysfunction in adults. It may cause muscle weakness, changes in glenohumeral kinematics, and instability in the shoulder internal and external rotator muscle groups and abductors. Patients may present a variety of symptoms, ranging from painless to severe shoulder pain and from normal function to severe dysfunction. It causes a decrease in the level of function in individuals, limitation in daily living activities, decreased quality of life and sleep problems. Various psychological factors, such as emotional or mental collapse and fear-avoidance behaviors, have been found to be associated with severe pain and disability in these patients. In response to emotional or physical injuries and traumas, fascia shortens, thickens, and stiffens. This situation causes pain and dysfunction. Conservative treatment is primarily preferred in the treatment of rotator cuff injury. In cases where there is no response to conservative treatment, surgery is used. Conservative treatment includes patient education, electrophysical agents, and exercise program. The exercise program includes scapular stabilization exercises, rotator cuff and shoulder area muscle strengthening exercises, range of motion exercises and stretching exercises. Additionally, the use of manual therapy techniques increases the effect of the treatment. Myofascial release technique, one of the manual therapy techniques, is a widely used therapy that involves low load and long-term mechanical forces to manipulate the myofascial complex, aiming to restore optimal length, reduce pain and improve function. With the myofascial release technique, proprioception is also increased. Considering the possible changes in the fascia, it is thought that the myofascial release technique may be useful in the conservative treatment program of individuals with rotator cuff injury. When the literature is examined, there is no study examining the effect of myofascial release technique on individuals with rotator cuff injury. The aim of this study is to investigate the long-term effects of myofascial release technique on proprioception, pain severity, shoulder range of motion, functional level, flexibility, and muscle strength in patients with rotator cuff injury.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of partial rotator cuff rupture
* Being between 18-65 years of age

Exclusion Criteria:

* Shoulder joint surgery
* Local steroid injection to the shoulder within the last 3 months
* Physiotherapy and rehabilitation within the last 3 months
* Cervical discopathy
* Severe shoulder osteoarthritis
* Upper extremity fracture or tumor
* Frozen shoulder
* Shoulder instability
* Thoracic outlet syndrome
* Neurological and mental problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Proprioception | Baseline
  Proprioception is the joint position sense. Shoulder flexion, abduction and external rotation proprioception were measured with a digital inclinometer. Deviations between the targeted angle and the angle performed by the patients were noted.
Proprioception | After four weeks of treatment
  Proprioception is the joint position sense. Shoulder flexion, abduction and external rotation proprioception were measured with a digital inclinometer. Deviations between the targeted angle and the angle performed by the patients were noted.
Pain severity | Baseline
  Pain is an unpleasant sensation and emotional experience. The severity of pain at rest and during activity was evaluated using visual analog scale. The starting point of the line indicated "no pain" and the end point "unbearable pain" using a 10 cm horizontal line.
Pain severity | After four weeks of treatment
  Pain is an unpleasant sensation and emotional experience. The severity of pain at rest and during activity was evaluated using visual analog scale. The starting point of the line indicated "no pain" and the end point "unbearable pain" using a 10 cm horizontal line.

SECONDARY OUTCOMES:
Range of motion | Baseline
  Range of motion is the measurement of movement. Active shoulder flexion, abduction, and internal and external rotation range of motion measurements were performed bilaterally with a universal goniometer in the supine position.
Range of motion | After four weeks of treatment
  Range of motion is the measurement of movement. Active shoulder flexion, abduction, and internal and external rotation range of motion measurements were performed bilaterally with a universal goniometer in the supine position.
Functional level | Baseline
  Functional level was assessed by Shoulder Pain and Disability Index (SPADI). SPADI consists of a total of 13 items, 5 of which determine the level of pain and 8 items that determine the level of disability.
Functional level | After four weeks of treatment
  Functional level was assessed by Shoulder Pain and Disability Index (SPADI). SPADI consists of a total of 13 items, 5 of which determine the level of pain and 8 items that determine the level of disability.
Flexibility | Baseline
  The ability to move muscles and joints through a full normal range of motion. Flexibility of the internal and external rotator muscles of the shoulder was measured with the patient in the sitting position. The measurement was made by recording the distance between the middle fingers of both hands with a tape measure.
Flexibility | After four weeks of treatment
  The ability to move muscles and joints through a full normal range of motion. Flexibility of the internal and external rotator muscles of the shoulder was measured with the patient in the sitting position. The measurement was made by recording the distance between the middle fingers of both hands with a tape measure.
Muscle strength | Baseline
  Shoulder flexor, abductor, and internal and external rotator muscle strength were measured bilaterally using a digital hand dynamometer. Measurements were made with the patient in the sitting position. For all measurements, patients were asked to respond to the resistance for 3 seconds. All of the procedures were repeated 3 times and 1 minute rest was given between sets.
Muscle strength | After four weeks of treatment
  Shoulder flexor, abductor, and internal and external rotator muscle strength were measured bilaterally using a digital hand dynamometer. Measurements were made with the patient in the sitting position. For all measurements, patients were asked to respond to the resistance for 3 seconds. All of the procedures were repeated 3 times and 1 minute rest was given between sets.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nho SJ, Yadav H, Shindle MK, Macgillivray JD. Rotator cuff degeneration: etiology and pathogenesis. Am J Sports Med. 2008 May;36(5):987-93. doi: 10.1177/0363546508317344. Epub 2008 Apr 15. PMID 18413681
- [Background] Celik MS, Sonmezer E, Acar M. Effectiveness of proprioceptive neuromuscular facilitation and myofascial release techniques in patients with subacromial impingement syndrome. Somatosens Mot Res. 2022 Jun-Dec;39(2-4):97-105. doi: 10.1080/08990220.2021.2018293. Epub 2022 Jan 7. PMID 34991428
- [Background] Gunes M, Yana M. Acute effects of thoracolumbar fascia release techniques on range of motion, proprioception, and muscular endurance in healthy young adults. J Bodyw Mov Ther. 2023 Jul;35:145-150. doi: 10.1016/j.jbmt.2023.04.063. Epub 2023 Apr 20. PMID 37330761